CLINICAL TRIAL: NCT04240327
Title: Marker Driven Selection of Patients for Prostate Biopsy and Management: The University of Miami MDSelect Protocol
Brief Title: Marker Driven Selection of Patients for Prostate Biopsy and Management
Acronym: MDSelect
Status: Active, not recruiting | Type: Observational
Sponsor: University of Miami (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Sanoj Punnen, MD, MAS, Associate Professor, University of Miami
Other Study IDs: 20190864; U01CA239141-01A1 (NIH); NCI-2020-05157 (Registry Identifier: NCI Clinical Trials Reporting Program (NCI CTRP))
Record Dates: First submitted 2020-01-20; First posted 2020-01-27 (Actual); Last update posted 2025-06-05 (Actual); Status verified 2025-06

CONDITIONS: PSA; Elevated PSA; Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Biopsy Tissue, blood and urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- GG2+ Prostate Cancer Risk: Participants at risk for Grade Group 2 (GG2+) prostate cancer. Participants will be followed for up to two years to rule out the presence of GG2+ prostate cancer

SUMMARY:
The purpose of this research study is to determine if the interpretation of multiparametric MRI (mpMRI) with an algorithm called habitat risk score (HRS) in combination with a panel of blood and urine biomarkers is more effective at detecting prostate cancer than standard of care interpretation of mpMRI with the Prostate Imaging Reporting and Data System (PIRADS).

ELIGIBILITY:
Inclusion Criteria:

1. Male participant, aged 40-85 years.
2. In good general health as evidenced by medical history.
3. Referred for a biopsy of the prostate for evaluation of prostate cancer due to elevated or increasing prostate-specific antigen (PSA) or an abnormal digital rectal exam (DRE).
4. Participant must agree to forego testosterone supplementation during the duration of the study due to unknown impacts on prostate cancer biomarkers.

Exclusion Criteria:

1. Previous or current history of prostate cancer or treatment for prostate cancer.
2. Previous history of pelvic radiation.
3. Known allergic reactions to MRI contrast or inability to undergo MRI due to renal toxicity.
4. Inability to undergo blood draw or biopsy of the prostate as per protocol.
5. Prior MRI guided biopsy of the prostate for prostate cancer evaluation.
6. Previous prostate biopsy or prostate procedure within 6 months of enrollment within the trial.
7. Standard contraindications to MRI, such as allergies to contrast die, renal toxicity, ferromagnetic metal in body/eye, pacemaker, defibrillator, other mechanical device, or extreme claustrophobia (medication with anti-anxiety agents, such as Ativan, may be attempted) will prevent eligibility and will be applied for all protocol-related MRIs.
8. Patients with impaired decision-making capacity.

Ages: 40 Years to 85 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study participants will be targeted for enrollment from a consecutive cohort of men who are referred to the University of Miami for prostate cancer evaluation and management, which includes internal and external physician referrals, most often due to an increased PSA, and/or abnormal digital rectal exam (DRE).
Sampling Method: Non-Probability Sample
Enrollment: 289 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Negative Predictive Value (NPV) for ruling out GG2+ prostate cancer via Habitat Risk Score (HRS) MRI Interpretation software combined with a panel of blood and urine biomarkers, versus via standard of care (SoC) MRI interpretation with PIRADS v2. | Up to 24 months
  The investigators will assess whether automated quantitative HRS MRI interpretation software combined with a panel of blood and urine biomarkers incrementally improves the negative predictive value for ruling out GG2+ cancer on prostate biopsy by 30% or more above standard of care (SoC) MRI interpretation with PIRADS v2.

SECONDARY OUTCOMES:
NPV for ruling out GG2+ prostate cancer via HRS MRI Interpretation software versus via SoC MRI interpretation with PIRADS v2 | Up to 24 months
  The investigators will assess whether automated quantitative HRS MRI interpretation software can incrementally improve the negative predictive value (NPV) for ruling out GG2+ cancer on prostate biopsy by 20% or more above SoC MRI interpretation with PIRADS v2.
NPV for ruling out GG2+ prostate cancer by a panel of blood and urine biomarkers versus via SoC MRI interpretation with PIRADS v2 | Up to 24 months
  The investigators will assess whether a panel of blood and urine biomarkers can incrementally improve the negative predictive value (NPV) for ruling out GG2+ cancer on prostate biopsy by 10% or more above SoC MRI interpretation with PIRADS v2.
NPV for ruling out clinically significant prostate cancer via HRS MRI interpretation software combined with a panel of blood and urine biomarkers versus via SoC MRI interpretation with PIRADS v2 | Up to 24 months
  The investigators will assess whether automated quantitative HRS MRI interpretation software combined with a panel of blood and urine biomarkers incrementally improves the negative predictive value for ruling out clinically significant prostate cancer (defined as any GG2+ cancer OR 50% or more cores of GG1 cancer) on prostate biopsy by 30% or more above standard of care MRI interpretation with PIRADS v2

CONTACTS AND LOCATIONS:
Overall Officials: Sanoj Punnen, MD, MAS, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No